CLINICAL TRIAL: NCT02592785
Title: An Open Label, Phase I Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Efficacy of BAY 1163877 in Japanese Subjects With Refractory, Locally Advanced or Metastatic Solid Tumors
Brief Title: Phase I Dose Escalation Study of BAY 1163877 (Rogaratinib) in Japanese Subjects With Refractory, Locally Advanced or Metastatic Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16958
Record Dates: First submitted 2015-10-29; First posted 2015-10-30 (Estimated); Last update posted 2018-04-18 (Actual); Status verified 2018-04

CONDITIONS: Neoplasms
MeSH Terms: conditions — Neoplasms | interventions — Rogaratinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- BAY1163877 (Experimental): Cohort 1: Safety, tolerability and PK of 600 mg dose given twice daily. Escalation to cohort 2 in case no safety relevant adverse event has been observed within 21 days after start of study treatment Cohort 2: Safety, tolerability and PK of 800 mg dose given twice daily
  Interventions: Drug: BAY1163877

INTERVENTIONS:
Drug: BAY1163877 — Cohort 1: Single dose 600 mg on day 1, no drug on day 2 and then twice daily administration of the same dose for the remaining 19 days of cycle 1. From cycle 2 onwards all subjects are continuously treated for 21 days per cycle with twice daily administration of the same dose.
  Cohort 2: Single dose 800 mg on day 1, no drug on day 2 and then twice daily administration of the same dose for the remaining 19 days of cycle 1. From cycle 2 onwards all subjects are continuously treated for 21 days per cycle with twice daily administration of the same dose.

SUMMARY:
Primary objectives of this study are to assess the safety and tolerability of BAY 1163877 in Japanese subjects with refractory, locally advanced or metastatic solid tumors and to characterize the PK of BAY 1163877

ELIGIBILITY:
Inclusion Criteria:

* Japanese males or female aged ≥ 20 years
* Histologically or cytologically confirmed refractory, locally advanced or metastatic solid tumors who are not candidates for standard therapy at discretion of investigator
* High FGFR expression levels based on archival or fresh tumor biopsy specimen analysis. Bladder cancer subjects with low overall FGFR expression levels can be included if activating FGFR3 mutations are confirmed.
* Subjects must have at least one measurable or evaluable lesion according to Response Evaluation Criteria in Solid Tumors, Version 1.1 (RECIST v1.1).
* Life expectancy of at least 3 months
* Recovery to National Cancer Institute's Common Terminology Criteria for Adverse Events, version 4.03 (CTCAE v4.03) Grade < 2 level or recovery to baseline preceding the prior treatment from any previous drug / procedure-related toxicity (subjects with persistent alopecia, anemia, and/or hypothyroidism can be included)
* Eastern Cooperative Oncology Group performance status (ECOG PS) of 0-2
* Adequate bone marrow, liver and renal function
* Prothrombin time-International normalized ratio (PT-INR) and activated partial thromboplastin time (APTT) ≤ 1.5 times ULN. Subjects being treated with anticoagulant, e.g. warfarin or heparin, will be allowed to participate provided no prior evidence of an underlying abnormality in these parameters exists

Exclusion Criteria:

* History or current condition of an uncontrolled cardiovascular disease including congestive heart failure New York Heart Association (NYHA) > Class 2, unstable angina (symptoms of angina at rest) or new-onset angina (within last 3 months) or myocardial infarction within past 6 months and cardiac arrhythmias requiring anti-arrhythmic therapy (beta-blockers or digoxin are permitted)
* Left ventricular ejection fraction (LVEF) < 50% as assessed by echocardiography performed
* Subjects with history and/or current evidence of endocrine alteration of calcium phosphate homeostasis (e.g. parathyroid disorder, history of parathyroidectomy, tumor lysis, tumoral calcinosis). Calcium (Ca) x (time) phosphate (PO4) should be < 70 mg²/dL².
* Current evidence of corneal disorder / keratopathy including but not limited to bullous / band keratopathy, corneal abrasion, inflammation / ulceration, keratoconjunctivitis etc. (to be confirmed by ophthalmologic examination). Pre-existing cataract is not an exclusion criterion.
* Moderate or severe hepatic impairment (subjects with Child-Pugh score B or C cannot be included.)
* Known human immunodeficiency virus (HIV) infection
* Subjects with an active hepatitis B and/or C infection requiring treatment
* Anticancer chemotherapy or immunotherapy during the study or within 5-half-lives of anticancer chemotherapy or immunotherapy before start of study treatment.
* Systolic blood pressure ≤ 110 and pulse rate ≥ 100/min, or diastolic blood pressure ≤ 70 mmHg and pulse rate ≥ 100/min
* Uncontrolled hypertension as indicated by a resting systolic BP ≥160 mmHg or diastolic BP ≥100 mmHg at screening

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2015-12-15 (Actual); Primary Completion 2017-02-05 (Actual); Study Completion 2017-12-06 (Actual)

PRIMARY OUTCOMES:
Number of an Treatment Emergent Adverse Event | Up to 35 days after the last study drug administration
Intensity of an Treatment Emergent Adverse Event graded using the NCI-CTCAE version 4.03 | Up tp 35 days after the last study drug administration
Maximum observed plasma concentration after single dose administration (Cmax) of BAY1163877 | On cycle 1, Day 1 to 3 (single-dose): Pre- dose, 0.5, 1, 2, 3, 4, 6, 8, 12, 24 and 48 hours post-dose
Cmax divided by dose (mg) per kg body weight (Cmax,norm) of BAY1163877 | On cycle 1, Day 1 to 3 (single-dose): Pre- dose, 0.5, 1, 2, 3, 4, 6, 8, 12, 24 and 48 hours post-dose
Cmax divided by dose (mg) (Cmax/D) of BAY1163877 | On cycle 1, Day 1 to 3 (single-dose): Pre- dose, 0.5, 1, 2, 3, 4, 6, 8, 12, 24 and 48 hours post-dose
Area under the plasma concentration vs time curve from zero to 12 hours p.a. after first-dose administration (AUC(0-12)) of BAY1163877 | On cycle 1, Day 1 to 3 (single-dose): Pre- dose, 0.5, 1, 2, 3, 4, 6, 8, 12 hours post-dose
AUC(0-12) divided by dose (mg) per kg body weight (AUC(0-12) norm) of BAY1163877 | On cycle 1, Day 1 to 3 (single-dose): Pre- dose, 0.5, 1, 2, 3, 4, 6, 8, 12 hours post-dose
AUC(0-12) divided by dose (mg) (AUC(0-12)/D) of BAY1163877 | On cycle 1, Day 1 to 3 (single-dose): Pre- dose, 0.5, 1, 2, 3, 4, 6, 8, 12 hours post-dose
AUC from time zero to the last data point > LLOQ (lower limit of quantification) of BAY1163877 (AUC(0-tlast)) | On cycle 1, Day 1 to 3 (single-dose): Pre- dose, 0.5, 1, 2, 3, 4, 6, 8, 12, 24 and 48 hours post-dose
AUC(0-tlast) divided by dose (mg) per kg body weight (AUC(0-tlast) norm) of BAY1163877 | On cycle 1, Day 1 to 3 (single-dose): Pre- dose, 0.5, 1, 2, 3, 4, 6, 8, 12, 24 and 48 hours post-dose
AUC(0-tlast) divided by dose (mg) (AUC(0-tlast)/D) of BAY1163877 | On cycle 1, Day 1 to 3 (single-dose): Pre- dose, 0.5, 1, 2, 3, 4, 6, 8, 12, 24 and 48 hours post-dose
AUC of BAY1163877 | On cycle 1, Day 1 to 3 (single-dose): Pre- dose, 0.5, 1, 2, 3, 4, 6, 8, 12, 24 and 48 hours post-dose
AUCnorm of BAY1163877 | On cycle 1, Day 1 to 3 (single-dose): Pre- dose, 0.5, 1, 2, 3, 4, 6, 8, 12, 24 and 48 hours post-dose
AUC/D of BAY1163877 | On cycle 1, Day 1 to 3 (single-dose): Pre- dose, 0.5, 1, 2, 3, 4, 6, 8, 12, 24 and 48 hours post-dose
Maximum Observed Drug Concentration in Plasma after multiple administrations (Cmax, md) of BAY1163877 | On cycle 1, Day 15 during multiple-dose: before morning dose and 0.5, 1, 2, 3, 4, 6, 8 and 12 hours post-dose
Cmax after multiple administrations divided by dose (mg) per kg body weight (Cmax,norm, md) of BAY1163877 | On cycle 1, Day 15 during multiple-dose: before morning dose and 0.5, 1, 2, 3, 4, 6, 8 and 12 hours post-dose
Cmax after multiple administrations divided by dose (mg) (Cmax/Dmd) of BAY1163877 | On cycle 1, Day 15 during multiple-dose: before morning dose and 0.5, 1, 2, 3, 4, 6, 8 and 12 hours post-dose
AUC(0-12) after multiple administrations (AUC(0-12)md) of BAY1163877 | On cycle 1, Day 15 during multiple-dose: before morning dose and 0.5, 1, 2, 3, 4, 6, 8 and 12 hours post-dose
AUC(0-12) after multiple administrations divided by dose (mg) per kg body weight (AUC(0-12)norm,md) of BAY1163877 | On cycle 1, Day 15 during multiple-dose: before morning dose and 0.5, 1, 2, 3, 4, 6, 8 and 12 hours post-dose
AUC(0-12) divided by dose (mg) after multiple administrations (AUC(0-12)/Dmd) of BAY1163877 | On cycle 1, Day 15 during multiple-dose: before morning dose and 0.5, 1, 2, 3, 4, 6, 8 and 12 hours post-dose
AUC(0-tlast)after multiple administrations (AUC(0-tlast)md) of BAY1163877 | On cycle 1, Day 15 during multiple-dose: before morning dose and 0.5, 1, 2, 3, 4, 6, 8 and 12 hours post-dose
AUC(0-tlast) after multiple administrations divided by dose (mg) per kg body weight (AUC(0-tlast) norm,md) of BAY1163877 | On cycle 1, Day 15 during multiple-dose: before morning dose and 0.5, 1, 2, 3, 4, 6, 8 and 12 hours post-dose
AUC(0-tlast) after multiple administrations divided by dose (mg) (AUC(0-tlast)/Dmd) of BAY1163877 | On cycle 1, Day 15 during multiple-dose: before morning dose and 0.5, 1, 2, 3, 4, 6, 8 and 12 hours post-dose

SECONDARY OUTCOMES:
Tumor response evaluation based on RECIST 1.1 | Screening, end of every second cycle (i.e., Cycle 2, 4, 6, 8,…)
FGF23 levels | Cycle 1 (Days 1 and 15)
  FGF 23: fibroblast growth factor 23
Phosphate levels | Cycle 1 (Days 1, 8, 15), Cycle 2 to 12 (Days 1, 8, 15), Cycle ≥13 (Days 1, 11), end of treatment
FGFR1/2/3 mRNA expression in tumor tissue to evaluate of biomarker status | At Screening visit

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (2):
- Japan (2):
  - Kashiwa, Chiba
  - Koto-ku, Tokyo